CLINICAL TRIAL: NCT03331159
Title: Evaluation of Fusion After Anterior Lumbar Interbody Fusion With a New Osteoinductive Bone Substitute Material: a First Randomized Clinical Trial
Brief Title: Evaluation of Fusion After ALIF With an Osteoinductive Material or With Homologus Bone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Mohammad ARAB MOTLAGH, MD, PhD, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NanoBone - ALIF
Record Dates: First submitted 2017-10-29; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Fusion of Spine, Lumbar Region
Keywords: Lumbar Fusion; Hydroxyapatite

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NanoBone (Experimental): The participants were treated with anterior lumbar interbody fusion (ALIF) with a new nanocrystalline hydroxyapatite embedded in a silica gel matrix (NH-SiO2)
  Interventions: Device: NanoBone
- Homologous bone (Active Comparator): The participants were treated with anterior lumbar interbody fusion (ALIF) with homologous bone
  Interventions: Device: Homologous Bone

INTERVENTIONS:
Device: NanoBone — Cage was filled with nanocrystalline hydroxyapatite embedded in a silica gel matrix
  Arms: NanoBone
Device: Homologous Bone — Cage was filled with homologous bone
  Arms: Homologous bone

SUMMARY:
The aim of this study was to determine whether instrumented anterior lumbar interbody Fusion with a new nanocrystalline hydroxyapatite embedded in a silica gel matrix (NH-SiO2) was associated with superior radiological and clinical outcomes at 12 months follow-up compared with instrumented ALIF with homologous bone

DETAILED DESCRIPTION:
This randomized clinical trial included two groups of 20 mature patients with mono- or multisegmental degenerative disease of the lumbar spine who were suitable to undergo mono- or bisegmental ALIF fusion at the level L4/L5 and L5/S1 with a carbon fiber reinforced polymer ALIF cage filled with either NH-SiO2 or homologous bone (HB). Patients were followed 12 months postoperatively. The primary aim was to compare postoperative disability as measured by the Oswestry Disability Index (ODI). Secondary aims were to compare postoperative radiographic outcomes and differences in pain and quality of life between these groups.

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain
* sensorimotor deficits
* radiculopathy and spinal claudication symptoms, all caused by degenerative changes in the lumbar spine, which were resistant to conservative pain therapy and / or physiotherapy

Exclusion Criteria:

* previous surgeries in the abdominal Region
* previous fusion surgery in the lumbar spine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2013-10-31 (Actual); Study Completion 2015-10-31 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | 12 months after surgery
  Postoperative disability as measured by the Oswestry Disability Index (ODI)

SECONDARY OUTCOMES:
Fusion rate | 12 months after surgery
  Postoperative radiographic Fusion rate

IPD SHARING:
Plan to Share IPD: No